CLINICAL TRIAL: NCT04697199
Title: The Adjunctive Effect of Probiotics to Non Surgical Treatment of Chronic Periodontitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ghadeer Khalil Elbagoory, Demonstrator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMP-02-18
Record Dates: First submitted 2020-12-31; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Chronic Periodontitis
Keywords: Chronic periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): patients received scaling and root planing using hand and ultrasonic instruments.
  Interventions: Procedure: Scaling and root planing
- Probiotic group (Active Comparator): patients received SRP and by using blunt syringe, subgingival delivery of 1ml of probiotic suspension was applied to these sites at baseline (immediately after SRP), one, two and four weeks. Periodontal dressing was applied after placement of the drug.
  After placement of the drug, patients were instructed to keep away from chewing hard or sticky food, brushing near the treated areas, or using any interdental aids for 24 hours.
  Interventions: Drug: Lactobacillus Reuteri Oral Drops; Procedure: Scaling and root planing

INTERVENTIONS:
Drug: Lactobacillus Reuteri Oral Drops — Subgingival delivery of probiotic suspension
  Other Names: Scaling and root planing
  Arms: Probiotic group
Procedure: Scaling and root planing — Scaling and root planing using hand and ultrasonic instruments

SUMMARY:
Evaluation of clinical and microbiological effect of lactobacillus reuteri probiotics.

DETAILED DESCRIPTION:
The present randomized controlled clinical trial was conducted to evaluate the effects of Lactobacillus reuteri-containing probiotic suspension as an adjunct to scaling and root planing (SRP).

Material and Methods: Twenty sites from twelve chronic periodontitis patients were recruited and monitored clinically and microbiologically at baseline, three, and six months after therapy for plaque index (PI), bleeding on probing (BOP), probing pocket depth (PPD) and clinical attachment level (CAL) and microbiologically or Porphyromonas gingivalis (P. gingivalis) load. Patients meeting the inclusion criteria were scheduled within one week for two sessions of SRP performed using ultrasonic scalers and hand instrumentation. After SRP, oral hygiene measures were reassured and then sites were randomly allocated to one of the two groups 10 sites each. group I (SRP only) and group II (SRP + probiotic). Group II received SRP and sub-gingival delivery of 1ml of probiotic L. reuteri suspension at baseline (immediately after SRP), one, two and four weeks using blunt syringe. Periodontal dressing was applied after placement of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with good systemic health.
2. Patients with moderate chronic periodontitis with attachment level ranging from 3-4 mm.
3. Optimal compliance as evidenced by no missed treatment appointments and positive attitude towards oral hygiene.
4. No gingival recession.

Exclusion Criteria:

1. Patients with history of antibiotic, anti-inflammatory drugs or periodontal therapy in the preceding 6 months.
2. Patients with risk factors (e.g. - smoking, uncontrolled diabetes, uncontrolled hypertension, pregnant or any other systemic disease which can alter the course of periodontal therapy).
3. Patients who are allergic to lactate products.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Change in Probing pocket depth | Baseline. 3 months. 6 months
  Individual acrylic stents were prepared to serve as the constant points to align the probe consistently and to reduce errors associated with probe placement. Probing pocket depth was assessed using a manual probe (UNC-15). The distance from the free gingival margin to the bottom of the pocket was recorded at six sites for each examined tooth. The probe was inserted in line with the long axis of the tooth and walked circumferentially around each surface of each tooth to detect and record the area of the deepest probe penetration. The mean probing pocket depth was obtained by summing the scores for the six sites and dividing it by six.

SECONDARY OUTCOMES:
Change in Plaque index | Baseline, 3 and 6 months
  This index distinguishes clearly between the severity and the location of soft debris aggregates.
Change in Bleeding on probing | Baseline, 3 and 6 months
  Bleeding on probing was performed through gentle probing of the orifice of the gingival crevice. If bleeding occurs within 10 seconds, the number of positive sites is recorded and then expressed as a percentage of the number of sites examined.
Change in Clinical attachment level | Baseline, 3 and 6 months
  The distance from cementoenamel junction to the bottom of the pocket was measured in the same way as described for probing

CONTACTS AND LOCATIONS:
Overall Officials: Elbagoory, Study Director — Tanta University
Locations (1):
- Ghadeer, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No